CLINICAL TRIAL: NCT01083095
Title: Establishment of a Sporozoite Challenge Model for Plasmodium Vivax in Human Volunteers
Acronym: ChallengeII
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Malaria Vaccine and Drug Development Center (Other)
Collaborators: Ministerio de la Protección Social, Colombia. (Unknown)
Responsible Party: Malaria Vaccine and Drug Development Center, Malaria Vaccine and Drug Development Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MVDC-2003-003; Reto II (Other: MVDC)
Record Dates: First submitted 2010-03-06; First posted 2010-03-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2006-12

CONDITIONS: Malaria, Vivax
Keywords: Malaria; Sporozoite; Challenge Model; Plasmodium vivax; Human Volunteers
MeSH Terms: conditions — Malaria, Vivax; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3 +/- 1 bite (Active Comparator): Volunteers were exposed to mosquito biting for 10 min
  Interventions: Biological: Sporozoite Challenge Model for Plasmodium vivax in Humans
- 6 +/- 1 bite (Active Comparator): Volunteers were exposed to mosquito biting for 10 min
  Interventions: Biological: Sporozoite Challenge Model for Plasmodium vivax in Humans
- 9 +/- 1 bite (Active Comparator): Volunteers were exposed to mosquito biting for 15 min
  Interventions: Biological: Sporozoite Challenge Model for Plasmodium vivax in Humans

INTERVENTIONS:
Biological: Sporozoite Challenge Model for Plasmodium vivax in Humans — Eighteen naïve volunteers were exposed to the bite of carrying P. vivax sporozoites. Volunteers were randomly allocated to 1 of 6 groups and exposed to different numbers of mosquito biting, for 10 min. After feeding, dissection of all mosquitoes exposed in the cage was performed, to confirm the presence of a blood meal in their midguts and sporozoites in their salivary glands. If a volunteer did not get the number of infective bites assigned for his/her group, he/she was allowed to be bitten for a new group of mosquitoes until a total of 3±1, 6±1, or 9±1 mosquito bites were achieved.
  Other Names: Controlled malaria vivax infection challenge

SUMMARY:
A clinical trial aimed to standardize a vivax sporozoite infection model in human volunteers was conducted at the Malaria Vaccine and Drug Development Center (MVDC) in collaboration with the Immunology Institute at Valle State University and the Fundación Clínica Valle del Lili (FCVL) in Cali, Colombia.

The primary objective was to determine if naïve human volunteers could be safely and reproducibly infected by the bite of An. albimanus mosquitoes carrying P. vivax sporozoites in their salivary glands and a secondary objective consisted in determining the minimal number of infected mosquitoes required to infect all volunteers, with a reproducible pre-patent period.

The trial was divided into two steps: Step A directed to obtain human blood infected with P.vivax parasite used to infect anopheles mosquitoes and Step B to produce P. vivax sporozoites in Anopheles mosquitoes to determine the dose response of naive human volunteers exposed to 3 +/- 1, 6 +/- 1 y 9 +/- 1 mosquitoes bites. A total of 15 samples of P. vivax infected donors were used to infect different batches of mosquitoes.

DETAILED DESCRIPTION:
Study design:

The study was a randomized open label clinical trial to establish a sporozoite challenge model for Plasmodium vivax in humans. The development and standardization of such a model will make it possible to evaluate the efficacy of candidate P. vivax vaccines in Phase 2a trials. The study is divided into two successive steps:

Step A Parasite Blood Donation: Volunteers were recruited passively from a group of patients who presented with active P. vivax infection and accepted to donate infected blood. Samples of P. vivax infected blood was collected and was screened for infectious diseases, according to standard blood bank procedures. Colonized Anopheles albimanus mosquitoes were fed with this blood using a Membrane Feeding Assay (MFA). Sixteen (16) days after, selected positive mosquito batches were used for step B.

Step B Challenge: After informed consent signature, a total of 18 healthy volunteers were randomly allocated to Groups 1, 2 and 3, of 6 volunteers each and were challenged with the bite of 3±1, 6±1 or 9±1 P. vivax infected mosquitoes. Volunteers were closely monitored post infection, and were treated as soon as blood infection becomes patent as ascertained by microscopic examination of thick blood smears (TBS). Comparison of three bite patterns was used to select the optimal number of P. vivax-infected mosquito bites needed to provide reliable and reproducible blood infection.

Infection was expected to occur in the first 30 days. After that time, if infection was not documented, antimalarial treatment was planned. Nevertheless all exposed volunteers presented malarial infection. Despite infection was expected before day 30, a 18 month follow-up was performed with to be sure no delay malaria infection presented without detection. So, the total duration of the study was 18 months.

Infection was determined by the detection of P. vivax parasites on TBS from volunteers included.

Eligibility criteria for Blood donors Step A were:

* Adult, male or female (18-60 years of age).
* Capacity to freely understand and sign an informed consent form of participation.
* TBS Positive for P.vivax but negative for all other malaria species.
* P.vivax gametocytemia > 0.2%.

Exclusion criteria

* Unable to provide free and willing written informed consent.
* Have or have had any illness or condition which, in the investigator's judgment, may substantially increase the risk associated with the blood donation.

Eligibility and exclusion criteria for Challenge is described below in this format.

Close monitoring of adverse events was performed, both by medical examination as by telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female adults (18- 50 years of age).
* Use of adequate contraceptive method from the initiation of the study until two months after sporozoite challenge for females.
* No plans to travel to a malaria endemic area during the course of the study and agree to not travel outside the study area from Day 7 to Day 23 post-challenge (the high risk period for becoming parasitemic).
* Reachable by phone during the entire study period
* Duffy positive phenotype

Exclusion Criteria:

* Are <18 or >49 years of age.
* Any female who is pregnant at serum positive B-HCG screening or who is nursing.
* Duffy negative phenotype.
* G-6-PD deficiency or any other hemoglobinopathy.
* Current or past infection with any species of malaria
* History of allergy to antimalarial drugs or immediate type hypersensitivity reactions to mosquito bites.
* Clinical or laboratory evidence of significant systemic disease, including hepatic, renal, cardiac, immunologic or hematological disease. Are HIV positive or have any other known immunodeficiency (including receiving immunosuppressive therapy or a history of splenectomy); are infected with hepatitis B or C virus; have a history of autoimmune disease (including inflammatory bowel disease, hemolytic anemia, autoimmune hepatitis, rheumatoid arthritis, lupus, etc.) or connective tissue disease or have any other serious underlying medical condition.
* Clinically significant laboratory abnormalities as determined by the Investigator(s).
* Plan to have surgery between enrollment and the end of the challenge follow-up.
* Have any other conditions that are determined by at least two concurring investigators that may interfere with the capacity to provide free and willing informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-01; Primary Completion 2005-03 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Percentage of infected naïve human volunteers after different number of infected mosquito biting | 30 days

SECONDARY OUTCOMES:
Minimal number of infected mosquitoes required to infect all volunteers with a reproducible prepatent period | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Socrates Herrera, MD, Principal Investigator — MVDC
Locations (1):
- Malaria Vaccine and Drug Testing Center, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Background] Clyde DF, Most H, McCarthy VC, Vanderberg JP. Immunization of man against sporozite-induced falciparum malaria. Am J Med Sci. 1973 Sep;266(3):169-77. doi: 10.1097/00000441-197309000-00002. No abstract available. PMID 4583408
- [Background] Good MF, Pombo D, Quakyi IA, Riley EM, Houghten RA, Menon A, Alling DW, Berzofsky JA, Miller LH. Human T-cell recognition of the circumsporozoite protein of Plasmodium falciparum: immunodominant T-cell domains map to the polymorphic regions of the molecule. Proc Natl Acad Sci U S A. 1988 Feb;85(4):1199-203. doi: 10.1073/pnas.85.4.1199. PMID 2448793
- [Background] Herrera MA, de Plata C, Gonzalez JM, Corradin G, Herrera S. Immunogenicity of multiple antigen peptides containing Plasmodium vivax CS epitopes in BALB/c mice. Mem Inst Oswaldo Cruz. 1994;89 Suppl 2:71-6. doi: 10.1590/s0074-02761994000600017. PMID 7565136
- [Result] Arevalo-Herrera M, Herrera S. Plasmodium vivax malaria vaccine development. Mol Immunol. 2001 Dec;38(6):443-55. doi: 10.1016/s0161-5890(01)00080-3. PMID 11741694
- [Result] Arevalo-Herrera M, Roggero MA, Gonzalez JM, Vergara J, Corradin G, Lopez JA, Herrera S. Mapping and comparison of the B-cell epitopes recognized on the Plasmodium vivax circumsporozoite protein by immune Colombians and immunized Aotus monkeys. Ann Trop Med Parasitol. 1998 Jul;92(5):539-51. PMID 9797827
- [Result] Baird JK, Tiwari T, Martin GJ, Tamminga CL, Prout TM, Tjaden J, Bravet PP, Rawlins S, Ferrel M, Carucci D, Hoffman SL. Chloroquine for the treatment of uncomplicated malaria in Guyana. Ann Trop Med Parasitol. 2002 Jun;96(4):339-48. doi: 10.1179/000349802125001023. PMID 12171615
- [Result] Blair S, Lopez ML, Pineros JG, Alvarez T, Tobon A, Carmona J. [Therapeutic efficacy of 3 treatment protocols for non-complicated Plasmodium falciparum malaria, Antioquia, Colombia, 2002]. Biomedica. 2003 Sep;23(3):318-27. Spanish. PMID 14582335
- [Result] Chotivanich K, Silamut K, Udomsangpetch R, Stepniewska KA, Pukrittayakamee S, Looareesuwan S, White NJ. Ex-vivo short-term culture and developmental assessment of Plasmodium vivax. Trans R Soc Trop Med Hyg. 2001 Nov-Dec;95(6):677-80. doi: 10.1016/s0035-9203(01)90113-0. PMID 11816444
- [Result] Chulay JD, Schneider I, Cosgriff TM, Hoffman SL, Ballou WR, Quakyi IA, Carter R, Trosper JH, Hockmeyer WT. Malaria transmitted to humans by mosquitoes infected from cultured Plasmodium falciparum. Am J Trop Med Hyg. 1986 Jan;35(1):66-8. doi: 10.4269/ajtmh.1986.35.66. PMID 3511753
- [Result] Church LW, Le TP, Bryan JP, Gordon DM, Edelman R, Fries L, Davis JR, Herrington DA, Clyde DF, Shmuklarsky MJ, Schneider I, McGovern TW, Chulay JD, Ballou WR, Hoffman SL. Clinical manifestations of Plasmodium falciparum malaria experimentally induced by mosquito challenge. J Infect Dis. 1997 Apr;175(4):915-20. doi: 10.1086/513990. PMID 9086149
- [Result] Clyde DF, McCarthy VC, Miller RM, Hornick RB. Specificity of protection of man immunized against sporozoite-induced falciparum malaria. Am J Med Sci. 1973 Dec;266(6):398-403. doi: 10.1097/00000441-197312000-00001. No abstract available. PMID 4590095
- [Result] Clyde DF. Immunization of man against falciparum and vivax malaria by use of attenuated sporozoites. Am J Trop Med Hyg. 1975 May;24(3):397-401. doi: 10.4269/ajtmh.1975.24.397. PMID 808142
- [Result] Clyde DF. Immunity to falciparum and vivax malaria induced by irradiated sporozoites: a review of the University of Maryland studies, 1971-75. Bull World Health Organ. 1990;68 Suppl(Suppl):9-12. PMID 2094597
- [Result] Collins WE, Jeffery GM. Primaquine resistance in Plasmodium vivax. Am J Trop Med Hyg. 1996 Sep;55(3):243-9. doi: 10.4269/ajtmh.1996.55.243. PMID 8842108
- [Result] Danis M. [Therapeutic advances against malaria in 2003]. Med Trop (Mars). 2003;63(3):267-70. French. PMID 14579464
- [Result] MCGREGOR IA, GILLES HM, WALTERS JH, DAVIES AH, PEARSON FA. Effects of heavy and repeated malarial infections on Gambian infants and children; effects of erythrocytic parasitization. Br Med J. 1956 Sep 22;2(4994):686-92. doi: 10.1136/bmj.2.4994.686. No abstract available. PMID 13356045
- [Result] Duarte EC, Pang LW, Ribeiro LC, Fontes CJ. Association of subtherapeutic dosages of a standard drug regimen with failures in preventing relapses of vivax malaria. Am J Trop Med Hyg. 2001 Nov;65(5):471-6. doi: 10.4269/ajtmh.2001.65.471. PMID 11716100
- [Result] Edelman R, Hoffman SL, Davis JR, Beier M, Sztein MB, Losonsky G, Herrington DA, Eddy HA, Hollingdale MR, Gordon DM, et al. Long-term persistence of sterile immunity in a volunteer immunized with X-irradiated Plasmodium falciparum sporozoites. J Infect Dis. 1993 Oct;168(4):1066-70. doi: 10.1093/infdis/168.4.1066. PMID 8376823
- [Result] Egan JE, Hoffman SL, Haynes JD, Sadoff JC, Schneider I, Grau GE, Hollingdale MR, Ballou WR, Gordon DM. Humoral immune responses in volunteers immunized with irradiated Plasmodium falciparum sporozoites. Am J Trop Med Hyg. 1993 Aug;49(2):166-73. doi: 10.4269/ajtmh.1993.49.166. PMID 8357078
- [Result] Fryauff DJ, Baird JK, Basri H, Sumawinata I, Purnomo, Richie TL, Ohrt CK, Mouzin E, Church CJ, Richards AL, et al. Randomised placebo-controlled trial of primaquine for prophylaxis of falciparum and vivax malaria. Lancet. 1995 Nov 4;346(8984):1190-3. doi: 10.1016/s0140-6736(95)92898-7. PMID 7475658
- [Result] Genton B, Corradin G. Malaria vaccines: from the laboratory to the field. Curr Drug Targets Immune Endocr Metabol Disord. 2002 Oct;2(3):255-67. doi: 10.2174/1568008023340613. PMID 12476490
- [Result] George FW 4th, Law JL, Rich KA, Martin WJ. Identification of a T-cell epitope on the circumsporozoite protein of Plasmodium vivax. Infect Immun. 1990 Feb;58(2):575-8. doi: 10.1128/iai.58.2.575-578.1990. PMID 1688828
- [Result] Glynn JR, Collins WE, Jeffery GM, Bradley DJ. Infecting dose and severity of falciparum malaria. Trans R Soc Trop Med Hyg. 1995 May-Jun;89(3):281-3. doi: 10.1016/0035-9203(95)90540-5. PMID 7660433
- [Result] Glynn JR, Bradley DJ. Inoculum size and severity of malaria induced with Plasmodium ovale. Acta Trop. 1995 Mar;59(1):65-70. doi: 10.1016/0001-706x(94)00078-f. PMID 7785527
- [Result] Glynn JR, Bradley DJ. Inoculum size, incubation period and severity of malaria. Analysis of data from malaria therapy records. Parasitology. 1995 Jan;110 ( Pt 1):7-19. doi: 10.1017/s0031182000080999. PMID 7845714
- [Result] Glynn JR. Infecting dose and severity of malaria: a literature review of induced malaria. J Trop Med Hyg. 1994 Oct;97(5):300-16. PMID 7932927
- [Result] Golenda CF, Li J, Rosenberg R. Continuous in vitro propagation of the malaria parasite Plasmodium vivax. Proc Natl Acad Sci U S A. 1997 Jun 24;94(13):6786-91. doi: 10.1073/pnas.94.13.6786. PMID 9192643
- See also: Related Info — http://www.inmuno.org